CLINICAL TRIAL: NCT00033553
Title: Induction/Concurrent Chemotherapy and Dose-Escalated Three Dimensional Thoracic Radiation for Patients With Stage III Non Small Cell Lung Cancer: A Randomized Phase II Study
Brief Title: Combination Chemotherapy and Computer-Planned Radiation Therapy in Treating Patients With Unresectable Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30105; U10CA031946 (NIH); CALGB-30105; CDR0000069300 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Carboplatin; Gemcitabine; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel + Carboplatin (Experimental): Paclitaxel and carboplatin induction (2 cycles)followed by chemotherapy with the addition of radiotherapy for 7 cycles
  Interventions: Drug: carboplatin; Drug: paclitaxel; Radiation: radiation therapy
- Gemcitabine + Carboplatin (Experimental): Gemcitabine and carboplatin induction (2cycles) followed by chemotherapy with the addition of radiotherapy for 7 cycles
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — Arm A: AUC=6 IV over 30 min for 2 cycles then AUC=2 IV over 30 min q wk for 7 wks Arm B: AUC=5 IV over 30 min for 2 cycles
Drug: gemcitabine hydrochloride — 1000 mg/sq m IV over 30 min days 1 & 8 repeat q 21 days for 2 cycles; then 35 mg/sq m IV over 30 min 2X wk for 7 wks
  Arms: Gemcitabine + Carboplatin
Drug: paclitaxel — 225 mg/sq m IV over 3 hrs q 21 days for 2 cycles, then 45 mg/sq m IV over 1 hr q wk for 7 wks
  Arms: Paclitaxel + Carboplatin
Radiation: radiation therapy — 3-D XRT 7400 cGy total after induction (during cycles 3-9)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Computer systems that allow doctors to create a 3-dimensional picture of the tumor to plan treatment may result in more effective radiation therapy. It is not yet known which chemotherapy and/or radiation therapy regimen is more effective in treating non-small cell lung cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of different combination chemotherapy regimens and 3-dimensional radiation therapy in treating patients who have unresectable stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall response rate, failure-free survival, and survival of patients with inoperable stage IIIA or IIIB non-small cell lung cancer treated with paclitaxel and carboplatin with concurrent 3-dimensional conformal radiotherapy (3-D XRT) vs gemcitabine and carboplatin with concurrent 3-D XRT.
* Compare the toxicity of these regimens in these patients.
* Compare the pattern of failure (locoregional vs distant failure) in patients treated with these regimens.
* Determine the feasibility of delivering 3-D XRT to patients in this multicenter study.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 2 courses. Patients then receive paclitaxel IV over 1 hour followed by carboplatin IV over 30 minutes once weekly and 3-dimensional conformal radiotherapy (3-D XRT) once daily 5 days a week. Treatment repeats weekly for 7 courses.
* Arm II: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 2 courses. Patients then receive gemcitabine IV over 30 minutes twice weekly and 3-D XRT as in arm I. Treatment repeats weekly for 7 courses.

In both arms, treatment continues in the absence of disease progression.

Patients are followed every 2 months for 2 years, every 4 months for 2 years, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 82 patients (41 per treatment arm) will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Squamous cell carcinoma
  * Adenocarcinoma, including bronchoalveolar cell carcinoma
  * Large cell anaplastic carcinoma, including giant and clear cell carcinoma
* Inoperable stage IIIA or IIIB disease
* No direct invasion of vertebral body

  * Tumors adjacent to a vertebral body without bone invasion allowed if all gross disease can be encompassed in radiotherapy boost field
* Contralateral mediastinal disease (N3) allowed if all gross disease can be encompassed in radiotherapy boost field
* No scalene, supraclavicular, or contralateral hilar node involvement
* Transudate, cytologically negative, non-bloody pleural effusion allowed if it can be encompassed in radiotherapy field

  * No exudative, bloody, or cytologically malignant pleural effusion
  * Evidence of pleural effusion by chest CT scan but not chest x-ray that is too small to tap allowed
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * The following are not considered measurable disease:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
    * Tumor lesions in a previously irradiated field

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* AST less than 2 times upper limit of normal

Renal:

* Creatinine clearance 20-130 mL/min for females
* Creatinine clearance 20-150 mL/min for males

Pulmonary:

* FEV1 at least 1.2 L

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other currently active malignancy (defined as completed prior therapy and considered to be at less than 30% risk of relapse) except non-melanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for NSCLC
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except steroids for adrenal failure or septic shock, hormones for non-disease-related conditions (e.g., insulin for diabetes), or glucocorticosteroids as antiemetics

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy for NSCLC

Surgery:

* At least 2 weeks since prior exploratory thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2002-03; Primary Completion 2006-09 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Response | 18 months post treatment
  Response is assessed as failure free survival

SECONDARY OUTCOMES:
Overall Survival | 6 years post treatment
Toxicity | 13 weeks
  Toxicity will be assessed during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Arthur William Blackstock, MD, Study Chair — Wake Forest University Health Sciences
Locations (74):
- United States (74):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Comprehensive Cancer Center at Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Socinski MA, Blackstock AW, Bogart JA, Wang X, Munley M, Rosenman J, Gu L, Masters GA, Ungaro P, Sleeper A, Green M, Miller AA, Vokes EE. Randomized phase II trial of induction chemotherapy followed by concurrent chemotherapy and dose-escalated thoracic conformal radiotherapy (74 Gy) in stage III non-small-cell lung cancer: CALGB 30105. J Clin Oncol. 2008 May 20;26(15):2457-63. doi: 10.1200/JCO.2007.14.7371. PMID 18487565
- [Result] Blackstock AW, Socinski MA, Bogart J, et al.: Induction (Ind) plus concurrent (Con) chemotherapy with high-dose (74 Gy) 3-dimensional (3-D) thoracic radiotherapy (TRT) in stage III non-small cell lung cancer (NSCLC): preliminary report of Cancer and Leukemia Group B (CALGB) 30105. [Abstract] J Clin Oncol 24 (Suppl 18): A-7042, 374s, 2006.
- [Result] Blackstock AW, Socinski MA, Gu L, et al.: Initial pulmonary toxicity evaluation of chemoradiotherapy (CRT) utilizing 74 Gy 3-dimensional (3-D) thoracic radiation in stage III non-small cell lung cancer (NSCLC): a Cancer and Leukemia Group B (CALGB) randomized phase II trial. [Abstract] J Clin Oncol 23 (Suppl 16): A-7060, 635s, 2005.